CLINICAL TRIAL: NCT07337603
Title: The Effect Of Trans-Anbdominal Pre-Peritoneal (TAPP) And Total Extra-Peritoneal (TEP) Procedures on Intraocular Pressure in Laparoscopıc Inguinal Hernia Repair :A Procspective Cohort Study
Brief Title: Intraocular Pressure in Laparoscopic Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Associate MD, Saglik Bilimleri Universitesi
Other Study IDs: EFSCH-2
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Groin Hernia; Intraocular Pressure
Keywords: TAPP procedure; TEP procedure; Groin Hernia; Intraocular Pressure
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAPP Group: Planned groin hernia patients who will operated with Transabdominal Preperitoneal technique
  Interventions: Other: Preoperative Intraocular Pressure; Other: Postoperative Intraocular Pressure
- TEP GRoup: Planned groin hernia patients who will operated with Trans Extra-Preperitoneal technique
  Interventions: Other: Preoperative Intraocular Pressure; Other: Postoperative Intraocular Pressure

INTERVENTIONS:
Other: Preoperative Intraocular Pressure — Preoperative Intraocular Pressure measurement for both eyes with Goldmann applanation tonometry before surgery
Other: Postoperative Intraocular Pressure — Postoperative first day's Intraocular Pressure measurement for both eyes with Goldmann applanation tonometry

SUMMARY:
Inguinal hernia is a common clinical condition, accounting for approximately 75% of abdominal wall hernias. The inguinal hernia surgery is one of the most common operations worldwide. The primary treatment for inguinal hernia is surgical options. In addition to the standard open surgical approach, the Lichtenstein technique, laparoscopic methods such as transabdominal preperitoneal (TAPP) and total extraperitoneal (TEP) approaches are currently the most commonly used surgical procedures.

Both methods result in less postoperative pain, seroma, chronic pain, hematoma, and wound infection compared to the Lichtenstein technique.

Many surgeons use the Trendelenburg position, approximately 30 to 45 degrees, when performing laparoscopic procedures. The advantage of the Trendelenburg position is that it allows for better visualization of the abdominal and pelvic organs and creates space for the operation. However, the Trendelenburg position also has some complications, such as increasing intraocular pressure. Also, in laparoscopic surgeries, pneumoperitoneum is created by introducing CO₂ gas into the abdomen. This increases intra-abdominal pressure, causing the diaphragm to be pushed upward and raising thoracic pressure. As a result, central venous pressure increases and intracranial venous return becomes difficult, which can lead to a temporary increase in intraocular pressure. Perioorbital swelling and venous congestion caused by prolonged surgery time and the position used can cause compartment syndrome in the orbital space and even lead to vision loss.

The current literature indicates that the increase in intra-abdominal pressure during laparoscopic surgery, the patient's position, and the surgery time can lead to an increase in intraocular pressure.

DETAILED DESCRIPTION:
Inguinal hernia is a common clinical condition, accounting for approximately 75% of abdominal wall hernias. It is more common in men than women, affecting approximately 25% of men and 2% of women throughout their lifetime. Due to its frequent occurrence, inguinal hernia surgery is one of the most common operations worldwide. The incidence of inguinal hernia shows a bimodal distribution, with the highest incidence occurring around the age of 5 and over 70. Two-thirds of these hernias are indirect hernias.

Many previous studies have identified several risk factors in its etiology, including advanced age, male gender, smoking, family history, conditions causing intra-abdominal pressure, and collagen connective tissue diseases.

The most fundamental point in diagnosing inguinal hernia is physical examination. Physical examination is the easiest and most accurate way to diagnose the hernia. However, while most inguinal hernias are diagnosed by physical examination, radiological examination may be necessary in cases where the body structure prevents physical examination. Radiological methods include ultrasonography, computed tomography and rarely magnetic resonance imaging.

The primary treatment for inguinal hernia is surgical options. In addition to the standard open surgical approach, the Lichtenstein technique, laparoscopic methods such as transabdominal preperitoneal (TAPP) and total extraperitoneal (TEP) approaches are currently the most commonly used surgical procedures.

The most frequently used laparoscopic treatment methods worldwide are TAPP and TEP procedures. In both methods, mesh is placed in the preperitoneal space, but in the TAPP technique, it is necessary to enter the abdominal cavity to place the mesh. In the TEP procedure, all procedures are performed without opening the peritoneal wall and without entering the abdomen.

While it is debated whether one procedure is superior to the other, there are discussions about their relative advantages and disadvantages. The most important advantage of the TEP procedure is that it is performed without entering the abdominal cavity; its disadvantage is that the surgeon performing the operation has to work in a narrower area. The advantages of the TAPP procedure are that it is a simpler technique, has a wider working area, and is suitable for bilateral evaluation. The disadvantage is the higher risk of intra-abdominal organ injury and intra-abdominal adhesions.

Both methods result in less postoperative pain, seroma, chronic pain, hematoma, and wound infection compared to the Lichtenstein technique.

Many surgeons use the Trendelenburg position, approximately 30 to 45 degrees, when performing laparoscopic procedures. The advantage of the Trendelenburg position is that it allows for better visualization of the abdominal and pelvic organs and creates space for the operation. However, the Trendelenburg position also has some complications, such as increasing intraocular pressure.

Also, in laparoscopic surgeries, pneumoperitoneum is created by introducing CO₂ gas into the abdomen. This increases intra-abdominal pressure, causing the diaphragm to be pushed upward and raising thoracic pressure. As a result, central venous pressure increases and intracranial venous return becomes difficult, which can lead to a temporary increase in intraocular pressure.

When the patient is placed in a head-down position, this return becomes even more difficult, and intraocular venous pressure increases even more. Similarly, prolonged surgery time can lead to increased hypoventilation and hypercapnia, which can cause choroidal congestion and increase intraocular pressure.

Perioorbital swelling and venous congestion caused by prolonged surgery time and the position used can cause compartment syndrome in the orbital space and even lead to vision loss.

The current literature indicates that the increase in intra-abdominal pressure during laparoscopic surgery, the patient's position, and the surgery time can lead to an increase in intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having been diagnosed with inguinal hernia
* Those wishing to participate in the study

Exclusion Criteria:

* Patients under 18 years of age
* Patients diagnosed with glaucoma
* Patients with rheumatological diseases (rheumatoid arthritis, SLE, etc.)
* Patients with chronic kidney and liver failure
* Patients who have undergone corneal transplantation
* Patients with malignancy
* Patients diagnosed with bilateral inguinal hernia
* Patients with ocular trauma
* Myopia or hyperopia exceeding three diopters
* Patients using systemic steroids
* Body Mass Index > 30 kg/m2
* Those who do not wish to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selecetive laparoscopic groin hernia repair patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
TAPP procedure effects intraocular pressure | Preooeratively and postoperative first day
  Preooeratively and postoperatively measured intraocular pressure with Goldmann's aplanasyon tonometry
TEP procedure effects intraocular pressure | Preooeratively and postoperative first day
  Preooeratively and postoperatively measured intraocular pressure with Goldmann's aplanasyon tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B Bozan, Professor, Study Director — Turkish Health Sciences University Elazig City Hospital
Locations (1):
- Elazig Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Primatesta P, Goldacre MJ. Inguinal hernia repair: incidence of elective and emergency surgery, readmission and mortality. Int J Epidemiol. 1996 Aug;25(4):835-9. doi: 10.1093/ije/25.4.835. PMID 8921464
- [Background] Rutkow IM. Epidemiologic, economic, and sociologic aspects of hernia surgery in the United States in the 1990s. Surg Clin North Am. 1998 Dec;78(6):941-51, v-vi. doi: 10.1016/S0039-6109(05)70363-7. PMID 9927978
- [Background] Lau H, Fang C, Yuen WK, Patil NG. Risk factors for inguinal hernia in adult males: a case-control study. Surgery. 2007 Feb;141(2):262-6. doi: 10.1016/j.surg.2006.04.014. Epub 2006 Jul 31. PMID 17263984
- [Background] Robinson A, Light D, Kasim A, Nice C. A systematic review and meta-analysis of the role of radiology in the diagnosis of occult inguinal hernia. Surg Endosc. 2013 Jan;27(1):11-8. doi: 10.1007/s00464-012-2412-3. Epub 2012 Jun 26. PMID 22733195
- [Background] Akhavan A, Gainsburg DM, Stock JA. Complications associated with patient positioning in urologic surgery. Urology. 2010 Dec;76(6):1309-16. doi: 10.1016/j.urology.2010.02.060. Epub 2010 May 23. PMID 20546878
- [Background] Kaur G, Sharma M, Kalra P, Purohit S, Chauhan K. Intraocular Pressure Changes during Laparoscopic Surgery in Trendelenburg Position in Patients Anesthetized with Propofol-based Total Intravenous Anesthesia Compared to Sevoflurane Anesthesia: A Comparative Study. Anesth Essays Res. 2018 Jan-Mar;12(1):67-72. doi: 10.4103/aer.AER_177_17. PMID 29628557
- [Background] Hoshikawa Y, Tsutsumi N, Ohkoshi K, Serizawa S, Hamada M, Inagaki K, Tsuzuki K, Koshimizu J, Echizen N, Fujitani S, Takahashi O, Deshpande GA. The effect of steep Trendelenburg positioning on intraocular pressure and visual function during robotic-assisted radical prostatectomy. Br J Ophthalmol. 2014 Mar;98(3):305-8. doi: 10.1136/bjophthalmol-2013-303536. Epub 2013 Sep 24. PMID 24064941
- [Background] Molloy BL. Implications for postoperative visual loss: steep trendelenburg position and effects on intraocular pressure. AANA J. 2011 Apr;79(2):115-21. PMID 21560974
- [Result] Aiolfi A, Cavalli M, Ferraro SD, Manfredini L, Bonitta G, Bruni PG, Bona D, Campanelli G. Treatment of Inguinal Hernia: Systematic Review and Updated Network Meta-analysis of Randomized Controlled Trials. Ann Surg. 2021 Dec 1;274(6):954-961. doi: 10.1097/SLA.0000000000004735. PMID 33427757
- [Result] Andresen K, Rosenberg J. Transabdominal pre-peritoneal (TAPP) versus totally extraperitoneal (TEP) laparoscopic techniques for inguinal hernia repair. Cochrane Database Syst Rev. 2024 Jul 4;7(7):CD004703. doi: 10.1002/14651858.CD004703.pub3. PMID 38963034
- [Result] Iossa A, Traumueller Tamagnini G, De Angelis F, Micalizzi A, Lelli G, Cavallaro G. TEP or TAPP: who, when, and how? Front Surg. 2024 Jul 15;11:1352196. doi: 10.3389/fsurg.2024.1352196. eCollection 2024. PMID 39077677
- [Result] Scheuermann U, Niebisch S, Lyros O, Jansen-Winkeln B, Gockel I. Transabdominal Preperitoneal (TAPP) versus Lichtenstein operation for primary inguinal hernia repair - A systematic review and meta-analysis of randomized controlled trials. BMC Surg. 2017 May 10;17(1):55. doi: 10.1186/s12893-017-0253-7. PMID 28490321
- [Result] Awad H, Santilli S, Ohr M, Roth A, Yan W, Fernandez S, Roth S, Patel V. The effects of steep trendelenburg positioning on intraocular pressure during robotic radical prostatectomy. Anesth Analg. 2009 Aug;109(2):473-8. doi: 10.1213/ane.0b013e3181a9098f. PMID 19608821